CLINICAL TRIAL: NCT01062880
Title: Neuropattern - Clinical Trial of a Psychobiological Stress Diagnostic Tool (Neuropattern - Erprobung Einer Psychobiologischen Stressdiagnostik)
Brief Title: Neuropattern - Assessment of a Translational Diagnostic Tool for Depression, Adjustment- and Somatoform-disorders
Acronym: Neuropattern
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Trier (Other)
Responsible Party: Prof. Dr. Dirk H. Hellhammer, University of Trier, Dept of Psychology, Div Clinical and Physiol Psychology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 961-38 62 61 / 891
Record Dates: First submitted 2010-02-03; First posted 2010-02-04 (Estimated); Last update posted 2010-02-04 (Estimated); Status verified 2009-10

CONDITIONS: Major Depression; Minor Depression; Somatoform Disorders; Adjustment Disorders
MeSH Terms: conditions — Depressive Disorder, Major; Somatoform Disorders; Adjustment Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: self-guided internet modules — Patients are assigned at random to either unspecific (n= 1000) or individualized (n=1000) self guided internet modules.

SUMMARY:
Neuropattern is a first translational tool in stress medicine. Neuropattern is a diagnostic tool, which can be applied by in- and outpatients and physicians to detect dysregulation in the stress response network. The physician provides anamnestic and anthropometric data, while the patient takes other measures at home, e.g. psychological, symptomatic, and biological data. Among the biological data are ECG measures for analyses of heart rate variability, and salivary cortisol measures before and after a dexamethasone challenge test. All data are analyzed in a central laboratory, which generates a written report for the physician, including a disease model, from which personalized recommendations for pharmacological and psychological treatments are derived. Neuropattern additionally offers individualized internet modules to inform the patient about the disease model and to teach him/her what he/she can do to improve his/her medical conditions. The current study applies Neuropattern in 2000 patients of family doctors, suffering from major depression, depressive episodes, adjustment disorders, and somatoform disorders. The patients receive either unspecific or individualized internet modules in a randomized order.

ELIGIBILITY:
Inclusion Criteria:

* native speakers
* ICD-F diagnoses 32, 33, 43.2, and 45

Exclusion Criteria:

* patients under glucocorticoid treatment
* patients taking antidepressants and anxiolytics
* patients under psychotherapeutic treatment
* pregnant women
* severe medical conditions
* mental retardation
* arrhythmia absoluta
* intolerance of dexamethasone

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2010-02; Primary Completion 2011-05 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Documentation and distribution of different endophenotypes (Neuropattern) in patients of family doctors suffering from depressive episodes, major depression, somatoform disorders, and adjustment disorders | 15 month

SECONDARY OUTCOMES:
Efficacy of Neuropattern diagnostics with respect to pharmacological treatments and internet based self-guided psychological modules | 1: start of diagnostic testing; 2: after 3 month; 3: after 6 month; 4: after 9 month

CONTACTS AND LOCATIONS:
Overall Officials: Dirk H Hellhammer, Professor, PhD, Principal Investigator — University of Trier, Dept. of Psychology
Locations (1):
- University of Trier, Department of Psychology, Clinical and Physiological Psychology, Trier, Germany

REFERENCES:
- [Background] Hellhammer, D.H., & Hellhammer, J. (Eds.). (2008). Stress: The Brain-Body Connection (Vol. 174). Basel: Karger.
- [Derived] Kumsta R, Kliegel D, Linden M, DeRijk R, de Kloet ER. Genetic variation of the mineralocorticoid receptor gene (MR, NR3C2) is associated with a conceptual endophenotype of "CRF-hypoactivity". Psychoneuroendocrinology. 2019 Jul;105:79-85. doi: 10.1016/j.psyneuen.2018.09.036. Epub 2018 Sep 27. PMID 30292651
- [Derived] Vogt D, Waeldin S, Hellhammer D, Meinlschmidt G. The role of early adversity and recent life stress in depression severity in an outpatient sample. J Psychiatr Res. 2016 Dec;83:61-70. doi: 10.1016/j.jpsychires.2016.08.007. Epub 2016 Aug 7. PMID 27566836